CLINICAL TRIAL: NCT02096471
Title: A Phase 2 Trial of the MEK Inhibitor PD-0325901 in Adolescents and Adults With NF1-Associated Morbid Plexiform Neurofibromas
Brief Title: MEK Inhibitor PD-0325901 Trial in Adolescents and Adults With NF1
Acronym: MEK Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Bruce Korf, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WI176190
Record Dates: First submitted 2014-03-12; First posted 2014-03-26 (Estimated); Results first posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2018-12

CONDITIONS: Neurofibromatosis Type 1 and Growing or Symptomatic, Inoperable PN
Keywords: Neurofibromatosis Type 1 (Neurofibromas); PD-0325901; Radiographic Response; Inoperable Plexiform Neurofibromas
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma | interventions — mirdametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Agent PD-0325901 (Experimental): The primary aim of the study will be to assess quantitative radiographic response in a target lesion. Subjects will receive PD-0325901 by mouth on a bid dosing schedule of 2 mg/m2/dose with a maximum dose of 4 mg bid. Each course is 4 weeks duration, and subjects will receive drug on a 3 week on/1 week off schedule. Subjects may receive additional courses beyond course 8 only if there is at least 15% reduction in volume of the target tumor. Subjects who have a 20% or greater reduction in target tumor volume at the end of 12 courses can continue on therapy for up to an additional year (maximum of 24 total courses). However, subjects who do not achieve at least 15% reduction in volume of the target tumor after 8 courses (~8 months) will be considered treatment failures and taken off study.
  Interventions: Drug: PD-0325901

INTERVENTIONS:
Drug: PD-0325901

SUMMARY:
This phase II open label study will evaluate adolescents (≥ 16 years of age) and adults with neurofibromatosis type-1 (NF1) and plexiform neurofibromas treated with the MEK inhibitor PD-0325901. The primary aim of the study will be to assess quantitative radiographic response in a target lesion. Subjects will receive PD-0325901 by mouth on a bid dosing schedule of 2 mg/m2/dose with a maximum dose of 4 mg bid. Each course is 4 weeks duration, and subjects will receive drug on a 3 week on/1 week off schedule. Subjects may receive additional courses beyond course 8 only if there is at least 15% reduction in volume of the target tumor. Subjects who have a 20% or greater reduction in target tumor volume at the end of 12 courses can continue on therapy for up to an additional year (maximum of 24 total courses). However, subjects who do not achieve at least 15% reduction in volume of the target tumor after 8 courses (~8 months) will be considered treatment failures and taken off study.

The Primary purpose of this protocol is to determine whether PD-0325901 results in objective radiographic responses based on volumetric MRI measurements in adolescents and adults with NF1 and growing or symptomatic inoperable PN.

There are several secondary aims of this protocol:

To evaluate the feasibility and toxicity of chronic PD-0325901 administration in this patient population

To estimate the objective response rate of up to 2 non-target plexiform neurofibromas to PD-0325901 by MRI

To characterize the pharmacokinetic profile of PD-0325901 when administered to this patient population

To evaluate quality of life and pain during treatment with PD-0325901

DETAILED DESCRIPTION:
This phase II open label study will evaluate adolescents (≥ 16 years of age) and adults with neurofibromatosis type-1 (NF1) and plexiform neurofibromas treated with the MEK inhibitor PD-0325901. The primary aim of the study will be to assess quantitative radiographic response in a target lesion. Subjects will receive PD-0325901 by mouth on a bid dosing schedule of 2 mg/m2/dose with a maximum dose of 4 mg bid. Each course is 4 weeks duration, and subjects will receive drug on a 3 week on/1 week off schedule. Subjects may receive additional courses beyond course 8 only if there is at least 15% reduction in volume of the target tumor. Subjects who have a 20% or greater reduction in target tumor volume at the end of 12 courses can continue on therapy for up to an additional year (maximum of 24 total courses). However, subjects who do not achieve at least 15% reduction in volume of the target tumor after 8 courses (~8 months) will be considered treatment failures and taken off study.

Subjects will have retinal screening performed before starting PD-0325901 and regularly while on study drug. Patients with glaucoma, intraocular pressure >21 mmHg, or any other significant abnormality (excluding chronic, stable ophthalmological findings secondary to Optic Pathway Glioma) on ophthalmic examination (performed by an ophthalmologist) will not be eligible. Patients who have received radiation or cytotoxic therapy within 4 weeks of study entry and patients who have received radiation to the orbit at any time previously, will not be eligible for the study. Patients with other concurrent severe and/or uncontrolled medical disease will also be excluded. In addition, pregnant women will not be eligible for enrollment and subjects of reproductive age will be required to practice birth control while on treatment.

Subjects entered on the trial will be carefully monitored for the development of PD-0325901 associated toxicities.

In all consenting subjects entered on this trial, a complete pharmacokinetic profile of PD-0325901 after administration will be evaluated during course 1. Involvement with this part of the study will be required.

Consenting subjects with dermal neurofibromas will have punch biopsies of dermal neurofibromas at two time points to determine if the PD-0325901 is affecting the biologic target. Involvement with this part of the study will be optional.

Since plexiform neurofibromas may significantly impact the lives of patients with NF1, this study will evaluate the effects of the disease and treatment with PD-0325901 on the quality of life (QOL) of adolescents and adults. Involvement in this part of the study will be required. The Pediatric Quality of Life Inventory (PedsQL) Neurofibromatosis Type 1 Module will be used to assess the QOL of subjects. The PedsQL NF1 Module is a self-reported disease-specific QOL scale developed for adolescents and adults with NF1. It assesses 16 domains of functioning including physical functioning, emotional functioning, social functioning, cognitive functioning, physical appearance, worry, pain and hurt, fatigue, and daily activities. Preliminary data collected on this scale indicates good reliability and validity in adults. The preliminary data in a small sample of adolescents also looks promising. Data collected from this trial may be used toward validating this instrument since no disease specific QOL measure for NF1 currently exists, but such a tool is critically needed. Pain will be assessed using the Numeric Rating Scale-11 (NRS-11), which is an 11-point self-report scale of pain intensity. In addition, the Brief Pain Inventory Pain Interference Scale is a 7-item self-report questionnaire that measures the extent to which pain interferes with daily functioning. Both of these brief measures have been recommended to assess different aspects of pain in clinical trials.

For subjects who respond to PD-0325901 (≥20% tumor volume reduction of target lesion by 12 courses), an MRI scan of the target lesion is requested (but not required) at 4 and 12 months after stopping drug (as long as the subject is still on protocol) in order to determine whether response is maintained post-therapy. These studies will not be requested from subjects who experience disease progression while on study drug.

Before the subject can be enrolled, the responsible institutional investigator must sign and date the completed eligibility checklist. The completed eligibility checklist should be faxed to the NF Operations Center to confirm eligibility prior to subject enrollment.

ELIGIBILITY:
Inclusion Criteria:

* All studies to determine eligibility must be performed within 2 weeks prior to enrollment unless otherwise indicated below. All clinical and laboratory data required for eligibility of a subject must be available in the subject's medical or research record.
* All subjects must have EITHER the clinical diagnosis of NF1 using the NIH Consensus Conference criteria OR have a constitutional NF1 mutation documented in a CLIA/CAP certified lab.
* Subjects must have plexiform neurofibroma(s) that are progressive OR are causing significant morbidity, such as (but not limited to) head and neck lesions that are compromising the airway or great vessels, brachial or lumbar plexus lesions that are causing nerve compression and loss of function, lesions causing major deformity (e.g., orbital lesions) or are significantly disfiguring lesions of the extremity that cause limb hypertrophy or loss of function, and painful lesions. Subjects with paraspinal plexiform neurofibromas will be eligible for this trial. Histologic confirmation of tumor is not necessary in the presence of consistent clinical and radiographic findings
* For subjects enrolled for tumor progression, progression is defined as:

  * Presence of new plexiform neurofibroma on MRI or CT (documented by comparison with prior MRI or CT), OR
  * A measurable increase in plexiform neurofibroma size (≥ 20% increase in the volume, or a ≥ 13% increase in the product of the two longest perpendicular diameters, or a ≥ 6% increase in the longest diameter) documented by comparison of two scans (MRI or CT) approximately one year or less prior to evaluation for this study.
* For subjects enrolled for a "major deformity" or "significantly disfiguring" tumor, eligible tumors will be limited to tumors of the head & neck or those on other areas of the body that are unable to be concealed by standard garments. In order to enroll a plexiform neurofibroma for these indications, the Study Chair or Co-Chair must be contacted to review subject eligibility prior to enrollment.
* Measurable disease: Subjects must have measurable plexiform neurofibroma(s) amenable to volumetric MRI analysis. The target lesion must be seen on at least 3 consecutive MRI slices and the field of view must contain the entire tumor of interest. Tumors must be at least 3 mL in volume (most PNs 3 cm in longest diameter will meet this criteria). If the tumor is <3 cm in longest diameter, the subject may still be eligible. Central review of the MRI of the target plexiform is required prior to enrollment to ensure that the tumor is measurable and amenable to volumetric analysis. After consenting, images will be sent for Central review
* Age: Subjects must be ≥ 16 years of age at the time of study entry.
* Durable Power of Attorney: Adults who are unable to provide informed consent will NOT be enrolled on this study.
* Performance Level: Karnofsky greater than or equal to 50% Note: Subjects who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Prior Therapy: Subjects are only eligible if complete resection of a plexiform neurofibroma with acceptable morbidity is not feasible, or if a subject with surgical option refuses surgery.
* Subjects who underwent surgery for a progressive plexiform neurofibroma will be eligible to enter the study after the surgery, provided the plexiform neurofibroma was incompletely resected and is evaluable by volumetric analysis.
* Subjects may have been previously treated for a plexiform neurofibroma or other tumor/malignancy, but must have fully recovered from the acute toxic effects of all prior chemotherapy or radiotherapy prior to entering this study.
* Myelosuppressive chemotherapy: Must not have received within 4 weeks of entry onto this study.
* Hematopoietic growth factors: At least 7 days since the completion of therapy with a growth factor that supports platelet, red or white cell number or function.
* Biologic (anti-neoplastic agent): At least 14 days since the completion of therapy with a biologic agent. These subjects must be discussed with the Study Chair on a case-by-case basis.
* Investigational Drugs: Subjects must not have received an investigational drug within 4 weeks.
* Steroids: Subjects with endocrine deficiencies are allowed to receive physiologic or stress doses of steroids if necessary.
* 6 months from involved field radiation to index plexiform neurofibroma(s); 6 weeks must have elapsed if subject has received radiation to areas outside index plexiform neurofibroma(s). Subjects who have received radiation to the orbit at any time are excluded.
* Surgery: At least 2 weeks since undergoing any major surgery and must be recovered from effects of surgery.
* Organ Function Requirements

  * Adequate Bone Marrow Function
  * Adequate Renal Function
  * Adequate Liver Function

Exclusion Criteria:

* Chronic treatment with systemic steroids or another immunosuppressive agent. Subjects with endocrine deficiencies are allowed to receive physiologic or stress doses of steroids if necessary.
* Evidence of an active optic glioma or other low-grade glioma, requiring treatment with chemotherapy or radiation therapy. Subjects not requiring treatment are eligible for this protocol.
* Patients with malignant glioma, malignant peripheral nerve sheath tumor, or other malignancy requiring treatment in the last 12 months.
* Subjects who have received radiation to the orbit at any time previously
* Subjects with glaucoma, intraocular pressure >21 mmHg, or any other significant abnormality on ophthalmic examination (performed by an ophthalmologist).
* Ophthalmological findings secondary to long-standing Optic Pathway Glioma such as optic nerve pallor or strabismus will NOT be considered significant for the purposes of the study.
* Tumor not able to be reliably evaluated by volumetric analysis.
* Other concurrent severe and/or uncontrolled medical disease, which could compromise participation in the study (e.g. uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, chronic liver or renal disease, active upper GI tract ulceration, congestive heart failure, etc.)
* Subjects who have an uncontrolled infection.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of PD-0325901 (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection). A nasogastric tube (NG tube) or gastric tube (G tube) is allowed.
* Women who are pregnant or breast feeding.
* Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method during the period they are receiving the study drug and for 3 months thereafter. Abstinence is an acceptable method of birth control. Women of childbearing potential will be given a pregnancy test within 7 days prior to administration of PD-0325901 and must have a negative urine or serum pregnancy test.
* History of noncompliance to medical regimens.
* Subjects unwilling to or unable to comply with the protocol, or who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
* Prior treatment with a MEK inhibitor of any kind

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-06; Primary Completion 2017-08-09 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Indiana Unversity, Indianapolis, Indiana
  - National Cancer Institute (NCI), Bethesda, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Washington University - St. Louis, St Louis, Missouri
  - New York University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Weiss BD, Wolters PL, Plotkin SR, Widemann BC, Tonsgard JH, Blakeley J, Allen JC, Schorry E, Korf B, Robison NJ, Goldman S, Vinks AA, Emoto C, Fukuda T, Robinson CT, Cutter G, Edwards L, Dombi E, Ratner N, Packer R, Fisher MJ. NF106: A Neurofibromatosis Clinical Trials Consortium Phase II Trial of the MEK Inhibitor Mirdametinib (PD-0325901) in Adolescents and Adults With NF1-Related Plexiform Neurofibromas. J Clin Oncol. 2021 Mar 1;39(7):797-806. doi: 10.1200/JCO.20.02220. Epub 2021 Jan 28. PMID 33507822

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study required at least 1 partial or complete response within the first 9 patients in order to complete recruitment.
Units Other Than Participants: Target Lesion
Groups:
- Agent PD-0325901: The primary aim of the study will be to assess quantitative radiographic response in a target lesion. Subjects will receive PD-0325901 by mouth on a bid dosing schedule of 2 mg/m2/dose with a maximum dose of 4 mg bid. Each course is 4 weeks duration, and subjects will receive drug on a 3 week on/1 week off schedule. Subjects may receive additional courses beyond course 8 only if there is at least 15% reduction in volume of the target tumor. Subjects who have a 20% or greater reduction in target tumor volume at the end of 12 courses can continue on therapy for up to an additional year (maximum of 24 total courses). However, subjects who do not achieve at least 15% reduction in volume of the target tumor after 8 courses (~8 months) will be considered treatment failures and taken off study.
  PD-0325901
Period: Overall Study
Arm/Group | Agent PD-0325901
Started | 19; 19 Target Lesion
Completed (This is a single group study and the units assigned data element is the target lesion.) | 6; 6 Target Lesion (Participants terminated the study if a partial response was not achieved and/or maintained.)
Not Completed | 13; 13 Target Lesion
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 7
Not completed — Withdrawal by Subject | 3
Not completed — Non-Compliant | 2

BASELINE CHARACTERISTICS:
Arm/Group | Agent PD-0325901
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.9 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 8
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19
MRI at Baseline [Count of Participants; unit: Participants] — All Eligible Patients
  Participants
    1 Target Number of Plexiform Neurofibromas | 17
    1 Target and non target Plexiform Neurofibromas | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With a 20% or More Change in Target Tumor Volume
Description: Response is assessed by the NCI-POB at the time that follow-up 3D-MRI scans are performed (after course 4, 8, 12, and then after completion of every 6 courses thereafter). For the purpose of determining the level of response (complete, partial, etc.) measurements from the follow-up scans are compared to the target lesion size in the pretreatment MRI scan using 3D data analysis.Complete Response (CR): A complete resolution of the target plexiform neurofibroma for ≥ 4 weeks Partial Response (PR): A ≥20% reduction in the volume of the target plexiform neurofibroma lesion for ≥4 weeks. Stable Disease (SD): A <20% increase, and < 20% decrease in the volume of the target plexiform neurofibroma lesion for ≥4 weeks.
  Progressive Disease (PD): A ≥ 20% increase in the volume (by 3D-MRI) of the target plexiform neurofibroma compared to the pretreatment volume..
Time Frame: baseline to 24 months
Population: All 19 participants enrolled equivalent to intention to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Agent PD-0325901
Number analyzed (Participants) | 19
Participants
  Complete response | 0
  Partial response | 8
  Stable response | 11
  Progressive Disease | 0

2. Secondary Outcome: Evaluable Participants Treated With PD-0325901
Description: Number of Evaluable Patients at 24 Months:
  Any subject with ≥ one dose of PD-0325901 and had a ≥ Grade 3 associated toxicity is evaluable for toxicity.
  In the absence of a ≥ Grade 3 toxicity, any subject who completed one full course of therapy is evaluable for toxicity.
  Evaluable For Response - Subjects who have completed at least two courses of therapy and have had their first follow-up MRI evaluation. Subjects who did not respond and are later found to have a target tumor other than a plexiform neurofibroma (e.g. malignant peripheral nerve sheath tumor) are not evaluable for response.
  Evaluable for Pharmacokinetics - Any subject who has at least 4 samples drawn for pharmacokinetics is evaluable for pharmacokinetics.
  Evaluable for Pharmacodynamics - Any subject who has a dermal neurofibroma biopsy for pharmacodynamics prior to starting therapy plus at least one other dermal neurofibroma biopsy is evaluable for
Time Frame: baseline to 24 months
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Agent PD-0325901
Number analyzed (Participants) | 19
Participants
  Evaluable | 8
  Failed to Achieve Comp/Partial Response | 11

3. Secondary Outcome: Toxicity of PD-0325901
Description: Number and Percent of Participants with AEs and SAEs
Time Frame: Baseline to 24 Months
Measure: Number; unit: participants
Arm/Group | Agent PD-0325901
Number analyzed (Participants) | 19
participants
  SAEs | 2
  AEs | 19

4. Secondary Outcome: The Objective Response Rate of up to 2 Non-Target Plexiform Neurofibromas to PD-0325901
Description: radiographic response based on volumetric MRI measurements of up to 2 Non Target Plexiform Neurofibromas classified as complete, partial, stable or progressive
Time Frame: Baseline to 24 Months
Population: All participants were evaluated and the two with non-Plexiform Neurofibromas were assessed.
Measure: Number; unit: participants
Arm/Group | Agent PD-0325901
Number analyzed (Participants) | 19
participants
  Complete response | 0
  Partial response | 0
  Stable response | 2
  Progressive Disease | 0

5. Secondary Outcome: Area Under the Curve for the Parent Compound
Description: Mean and Standard Deviation AUC Estimates of the levels of PD-0325901 over 12-Hours for both the Parent and Metabolite Compound, based on samples at Pre-dose, .5 Hr. Post dose, 1.0 Hr.Post dose, 2.0 Hr.Post dose, 3.0 Hr. Post dose, 4.0 Hr.Post dose, 6.0 Hr. Post dose, 8.0 Hr. Post dose, 10.0-12.0 Hr. Post dose.
Time Frame: Day 1; Course 1
Population: 18 of the 19 participants had PK samples drawn.
Measure: Mean (Standard Deviation); unit: ng/mL*hr/(mg/m^2Parent)
Arm/Group | Agent PD-0325901
Number analyzed (Participants) | 18
ng/mL*hr/(mg/m^2Parent) | 219.1 (41.4)

6. Secondary Outcome: Quality of Life Using the Pain Subscale of the NRS-11 and PedsQL™ NF1 for Subjects Receiving PD-0325901 Using Age-based Assessments
Description: The PedsQL™ NF1 Module asks how much of a problem each item has been during the past one month. A 5-point response scale: 0= never a problem...4= almost always a problem). Items are reverse scored and linearly transformed to a scale of 0-100 Higher scores = better HRQOL. The total scale score is the sum of items divided by the number answered. Subscale scores are computed similarly. If more than 50% of the items in the scale are missing, the scale score is not computed. The Numerical Rating Scale-11 (NRS-11) is a self-report segmented 11-point numeric scale that assesses pain intensity with 0 representing "no pain" at the right end of the line and 10 representing "worst pain you can imagine". The Brief Pain Inventory (BPI)-Pain Interference Scale is a 7-item self-report questionnaire asking (general activity, mood, walking, normal work, relations with other people, sleep, and enjoyment of life) in the past week with 0 = no interference and 10 = completely interferes.
Time Frame: Baseline to 12 Months
Population: NRS-11 are on a scale of 0-10 with 0 being no pain, higher scores are greater intensity. BPI pain interference scale yields a total score (each item 0-10 and total score=mean all items) higher scores are more pain interference.Remaining items are initially a 5-point Likert scale (0-4) and transformed to a 0-100 scale with higher scores better QOL.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Agent PD-0325901
Number analyzed (Participants) | 19
score on a scale
  Overall Tumor Pain Change (Baseline - 12 mo.) | 1.38 (0.84)
  Most Important Tumor Pain (Baseline - 12 mo.) | 2.10 (0.80)
  Brief Pain Inventory (Baseline - 12 mo.) | 0.89 (0.66)
  Total Functioning (Baseline - 12 mo.) | -3.77 (3.60)
  Physical Functioning (Baseline - 12 mo.) | -3.55 (6.87)
  Pain and Hurt (Baseline - 12 mo.) | -13.06 (8.29)
  Movement and Balance (Baseline - 12 mo.) | -12.98 (6.35)
  Daily Activities (Baseline - 12 mo.) | 6.66 (5.05)
  Emotional Functioning (Baseline - 12 mo.) | -2.34 (6.46)
  Social Functioning (Baseline - 12 mo.) | -6.24 (6.79)
  Cognitive Functioning (Baseline - 12 mo.) | -0.17 (6.37)
  Communication Functioning (Baseline - 12 mo.) | 0.68 (7.99)
  Worry (Baseline - 12 mo.) | -10.97 (8.16)
  Paresthesias (Baseline - 12 mo.) | -3.74 (6.58)
  Skin Irritation (Baseline - 12 mo.) | -4.21 (5.51)
  Sensation (Baseline - 12 mo.) | -6.27 (5.72)
  Fatigue (Baseline - 12 mo.) | -0.71 (8.52)
  Treatment Anxiety (Baseline - 12 mo.) | -1.07 (7.53)
Statistical Analysis 1: Comparison: Agent PD-0325901; Single group change from baseline; Test type: Superiority — Single group study. Change in Pain from Baseline amongst those with a tumor response; p = 0.11, t-test, 2 sided; Descriptive analysis only; Mean Difference (Final Values) = 1.38, Standard Error of Mean 0.84
Statistical Analysis 2: Comparison: Agent PD-0325901; Single Group Change from Baseline; Test type: Superiority — Single Group Study. Change in Pain from Baseline amongst those with a Tumor Response; p = 0.01, t-test, 2 sided; Descriptive Analysis Only; Mean Difference (Final Values) = 2.10, Standard Error of Mean 0.80
Statistical Analysis 3: Comparison: Agent PD-0325901; Single Group Change from Baseline; Test type: Superiority — Single Group Study. Change in Pain from Baseline amongst those with a Tumor Response; p = 0.18, t-test, 2 sided; Descriptive Analysis Only; Mean Difference (Final Values) = 0.89, Standard Error of Mean 0.66
Statistical Analysis 4: Comparison: Agent PD-0325901; Single Group Change from Baseline; Test type: Superiority — Single Group Study. Change in Quality of Life (QOL) from Baseline amongst those with a Tumor Response; p = 0.30, t-test, 2 sided; Descriptive Analysis Only; Mean Difference (Final Values) = -3.77, Standard Error of Mean 3.60
Statistical Analysis 5: Comparison: Agent PD-0325901; Single Group Change from Baseline; Test type: Superiority — Single Group Study Change in Quality of Life from Baseline amongst those with a Tumor Response; p = 0.61, t-test, 2 sided; Descriptive Analysis Only; Mean Difference (Final Values) = -3.55, Standard Error of Mean 6.87
Statistical Analysis 6: Comparison: Agent PD-0325901; Single Group Change from Baseline; Test type: Superiority — Single Group Study Change in Baseline amongst those with a Tumor Response; p = 0.12, t-test, 2 sided; Descriptive Analysis Only; Mean Difference (Final Values) = -13.06, Standard Error of Mean 8.29
Statistical Analysis 7: Comparison: Agent PD-0325901; Single Group Change from Baseline; Test type: Superiority — Single Group Study. Change in Quality of Life from Baseline amongst those with a Tumor Response; p = 0.05, t-test, 2 sided; Descriptive Analysis Only; Mean Difference (Final Values) = -12.98, Standard Error of Mean 6.35
Statistical Analysis 8: Comparison: Agent PD-0325901; Single Group Change from Baseline; Test type: Superiority — Single Group Study. Change in Quality of Life from Baseline amongst those with a Tumor Response; p = 0.19, t-test, 2 sided; Descriptive Analysis Only; Mean Difference (Final Values) = 6.66, Standard Error of Mean 5.05
Statistical Analysis 9: Comparison: Agent PD-0325901; Single Group Change from Baseline; Test type: Superiority — Single Group Study. Change in Quality of Life from Baseline amongst those with a Tumor Response; p = 0.72, t-test, 2 sided; Descriptive Analysis Only; Mean Difference (Final Values) = -2.34, Standard Error of Mean 6.46
Statistical Analysis 10: Comparison: Agent PD-0325901; Single Group Change from Baseline; Test type: Superiority — Single Group Study. Change in Quality of Life from Baseline amongst those with a Tumor Response; p = 0.36, t-test, 2 sided; Descriptive Analysis Only; Mean Difference (Final Values) = -6.24, Standard Error of Mean 6.74
Statistical Analysis 11: Comparison: Agent PD-0325901; Single Group Change from Baseline; Test type: Superiority — Single Group Study. Change in Quality of Life from Baseline amongst those with a Tumor Response; p = 0.98, t-test, 2 sided; Descriptive Analysis Only; Mean Difference (Final Values) = -0.17, Standard Error of Mean 6.37
Statistical Analysis 12: Comparison: Agent PD-0325901; Single Group Change from Baseline; Test type: Superiority — Single Group Study. change in Quality of Life from Baseline amongst those with a Tumor Response; p = 0.93, t-test, 2 sided; Descriptive Analysis Only; Mean Difference (Final Values) = 0.68, Standard Error of Mean 7.99
Statistical Analysis 13: Comparison: Agent PD-0325901; Single Group Change from Baseline; Test type: Superiority — Single Group Study. Change in Quality of Life from Baseline amongst those with a Tumor Response; p = 0.19, t-test, 2 sided; Descriptive Analysis Only; Mean Difference (Final Values) = -10.97, Standard Error of Mean 8.16
Statistical Analysis 14: Comparison: Agent PD-0325901; Single Group Change from Baseline; Test type: Superiority — Single Group Study. Change in Quality of Life from Baseline amongst those with a Tumor Response; p = 0.57, t-test, 2 sided; Descriptive Analysis Only; Mean Difference (Final Values) = -3.74, Standard Error of Mean 6.58
Statistical Analysis 15: Comparison: Agent PD-0325901; Single Group Change from Baseline; Test type: Superiority — Single Group Study. Change in Quality of Life from Baseline amongst those with a Tumor Response; p = 0.45, t-test, 2 sided; Descriptive Analysis Only; Mean Difference (Final Values) = -4.21, Standard Error of Mean 5.51
Statistical Analysis 16: Comparison: Agent PD-0325901; Single Group Change from Baseline; Test type: Superiority — Single Group Study. Change in Quality of Life from Baseline amongst those with a Tumor Response; p = 0.28, t-test, 2 sided; Descriptive Analysis Only; Mean Difference (Final Values) = -6.27, Standard Error of Mean 5.72
Statistical Analysis 17: Comparison: Agent PD-0325901; Single Group Change from Baseline; Test type: Superiority — Single Group Study. Change in Quality of Life from Baseline amongst those with a Tumor Response; p = 0.93, t-test, 2 sided; Descriptive Analysis Only; Mean Difference (Final Values) = -0.71, Standard Error of Mean 8.52
Statistical Analysis 18: Comparison: Agent PD-0325901; Single Group Change from Baseline; Test type: Superiority — Single Group Study. Change in Quality of Life from Baseline amongst those with a Tumor Response; p = 0.89, t-test, 2 sided; Descriptive Analysis Only; Mean Difference (Final Values) = -1.07, Standard Error of Mean 7.53

7. Secondary Outcome: Area Under the Curve for the Metabolite Compound
Description: Mean 12-Hour AUC Estimates of the Parent and Metabolite Compound, based on samples at Pre-dose, .5 Hr. Post dose, 1.0 Hr.Post dose, 2.0 Hr.Post dose, 3.0 Hr. Post dose, 4.0 Hr.Post dose, 6.0 Hr. Post dose, 8.0 Hr. Post dose, 10.0-12.0 Hr. Post dose.
Time Frame: Day 1; Course 1
Population: 18 of the 19 participants had PK samples collected and the metabolite compound AUC was computed and summarized.
Measure: Mean (Standard Deviation); unit: ng/mL*hr/(mg/m^2 Metabolite)
Arm/Group | Agent PD-0325901
Number analyzed (Participants) | 18
ng/mL*hr/(mg/m^2 Metabolite) | 91.1 (49.5)

8. Secondary Outcome: Mean Half-Life for the PD-0325901 Concentrations
Description: Half life Estimates of PD-0325901 of the Parent and Metabolite Compound, based on samples at Pre-dose, .5 Hr. Post dose, 1.0 Hr.Post dose, 2.0 Hr.Post dose, 3.0 Hr. Post dose, 4.0 Hr.Post dose, 6.0 Hr. Post dose, 8.0 Hr. Post dose, 10.0-12.0 Hr. Post dose.
Time Frame: Day 1; Course 1
Population: 18 of the 19 participants had PK samples collected and the metabolite compound AUC was computed and summarized.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Agent PD-0325901
Number analyzed (Participants) | 18
hours | 6.1 (3.5)

ADVERSE EVENTS:
Time Frame: Baseline to 24 Months
Arm/Group | Agent PD-0325901
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Agent PD-0325901 (N=19)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pregnancy, puerperium and perinatal conditions, other (Pregnancy, puerperium and perinatal conditions) | 1 (1) — Male subject reported noncompliance with contraception and fathered a pregnancy.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Agent PD-0325901 (N=19)
Anemia (Blood and lymphatic system disorders) | 3
Hemolysis (Blood and lymphatic system disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Eye Disorder - Other, Pigment Changes (Eye disorders) | 1
Eye Disorder - Other, Subconjunctival Hemmorrhage of the Eye (Eye disorders) | 1
Eye Disorders - Other, Choroidal Space Macular (Eye disorders) | 1
Eye Disorders - Other, Nuclear Lens Opacification (Eye disorders) | 1
Eye Disorders - Other, Optic Nerve Drusen (Eye disorders) | 1
Eye Pain (Eye disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 3
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 6
Dry Mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, Blood in Stool (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, Duodenitis (Gastrointestinal disorders) | 1
Gastroparesis (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 12
Oral Pain (Gastrointestinal disorders) | 1
Rectal hemmorrhage (Gastrointestinal disorders) | 1
Vomitting (Gastrointestinal disorders) | 7
Chills (General disorders) | 1
Edema Face (General disorders) | 1
Edema Limbs (General disorders) | 2
Fatigue (General disorders) | 11
Flu-like Symptoms (General disorders) | 3
Localized Edema (General disorders) | 1
Pain (General disorders) | 2
Conjunctivitis Infective (Infections and infestations) | 1
Mucosal Infection (Infections and infestations) | 1
Paronychia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Tooth Infection (Infections and infestations) | 1
Upper Respiratory Infection (Infections and infestations) | 3
Alkaline Phosphatase Increased (Investigations) | 1
Aspartate Aminotransferase Increased (Investigations) | 2
Blood Bilirubin Increased (Investigations) | 1
CPK Increased (Investigations) | 6
Creatinine Increased (Investigations) | 1
Hemoglobin Increased (Investigations) | 1
Hiatal Hernia (Investigations) | 1
Indigestion (Investigations) | 1
Investigations - Other, Total Protein Serum High (Investigations) | 1
Lymphocyte Count Decreased (Investigations) | 2
Lymphocyte Count Increased (Investigations) | 1
Neutrophil Count Decreased (Investigations) | 1
Platelet Count Decreased (Investigations) | 2
Weight Gain (Investigations) | 3
White Blood Cell Count Decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypernatermia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hyerkalemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Fibrosis Deep Connective Tissue (Musculoskeletal and connective tissue disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorders - Other, Hip Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4
Neoplasms benign, malignant and unspecified (inc cysts and polyps) - Other, Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 8
Movements involuntary (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 2
Spasticity (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Irregular menstruation (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - other, breakthrough bleeding (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Alpecia (Skin and subcutaneous tissue disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash maculopapular (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 18
Rash pustular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, Bleeding and oozing from ear (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, Erythema hallux (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, Erythema (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, Hemangiomas (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, Oily Skin (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, Pustular Dermatosis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2
Vascular disorder - Other, Hot Flashes (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
None to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT02096471/Prot_SAP_000.pdf